CLINICAL TRIAL: NCT02195895
Title: 12 Month Open-Label Extension Study of the Effect of Alendronate on Bone in People With Chronic SCI Previously Treated With Teriparatide
Brief Title: Effect of Alendronate on Bone in People With Chronic Spinal Cord Injury (SCI) Previously Treated With Teriparatide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00083759
Record Dates: First submitted 2014-07-14; First posted 2014-07-21 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injury; Bone Loss; Osteoporosis
Keywords: Teriparatide; Alendronate; Alendronic Acid; Osteoporosis; Bone Fracture; Bone Loss; Spinal Cord Injury; Bone Diseases; Metabolic Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Nervous System; Wounds and Injuries; Bone Density Conservation Agents; Physiological Effects of Drugs; Pharmacologic Actions
MeSH Terms: conditions — Spinal Cord Injuries; Bone Diseases, Metabolic; Osteoporosis; Fractures, Bone; Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Wounds and Injuries | interventions — Alendronate; Calcium; Calcium Carbonate; Antacids; Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alendronate, Calcium, Vitamin D (Experimental): Drug: Weekly oral alendronate 70 mg for 12 months
  Supplements: 1000 mg Calcium and 1000 IU Vitamin D daily for 12 months
  Interventions: Drug: Alendronate; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Alendronate — Weekly oral alendronate 70 mg for 12 months
  Other Names: Alendronic acid; Fosamax
Dietary Supplement: Calcium — Daily oral 1000 mg Calcium
  Other Names: Calcium carbonate; Antacid
Dietary Supplement: Vitamin D — Daily oral 1000 IU
  Other Names: Vitamin D3; Cholecalciferol

SUMMARY:
The purpose of this study is to determine if a year of alendronate treatment will maintain or increase bone mass density (BMD) compared to baseline BMD values in people with chronic spinal cord injury (SCI).

This study will also investigate 1) if alendronate therapy will increase bone strength in people with chronic SCI, 2) the number of participants with adverse events from alendronate, and 3) the effects of alendronate on serum markers of bone metabolism.

DETAILED DESCRIPTION:
This extension study will enroll individuals who have completed treatment in the parent protocol "Effect of Teriparatide, Vibration and the Combination on Bone Mass and Bone Architecture in Chronic Spinal Cord Injury" or in the teriparatide extension protocol. This study will allow those individuals who previously received teriparatide to be treated for a year with alendronate to maintain any bone they may have gained and to possibly increase bone mass further. Termination of teriparatide is followed by bone loss if anti-resorptive therapy is not initiated, so this approach is optimal for continued treatment of the current group of participants.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in protocol "Effect of Teriparatide, Vibration and the Combination on Bone Mass and Bone Architecture in Chronic Spinal Cord Injury", (NCT01225055).
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Individual with renal insufficiency (calculated creatinine clearance < 30 ml/min).
* Individuals who are not able to sit or stand upright for at least 30 minutes after taking their medication.
* Individuals with poor dental hygiene.
* Individuals with esophageal abnormalities.
* Individuals who are not able to tolerate alendronate treatment.
* Individuals who will not be able to return for all study visits.
* Patients may not be receiving any other investigational agents.
* Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alendronate, Calcium, Vitamin D: Drug: Weekly oral alendronate 70 mg for 12 months
  Supplements: Calcium and Vitamin D daily for 12 months
  Alendronate: Weekly oral alendronate 70 mg for 12 months
  Calcium: Daily Oral 1000 mg
  Vitamin D: Daily Oral 1000 IU
Period: Overall Study
Arm/Group | Alendronate, Calcium, Vitamin D
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 43.89 [23.13 to 68.05]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
American Spinal Injury Association (ASIA) Impairment Scale [Count of Participants; unit: Participants] — ASIA impairment scale describes a person's functional impairment as a result of their spinal cord injury.
  A = Complete. No motor or sensory function in the lowest sacral spine segment (S4-5).
  B = Sensory Incomplete. Sensory function below the neurological level of injury (NLI) and in S4-S5, no motor function below NLI.
  C = Motor Incomplete. Motor function is preserved below NLI and more than half of the key muscle groups below NLI have a muscle grade < 3.
  D = Motor Incomplete. Motor function is preserved below NLI and at least half of the key muscle groups below NLI have a muscle grade 3.
  Participants
    ASIA A (Complete Injury) | 12
    ASIA B (Sensory Incomplete Injury) | 1
    ASIA C (Motor Incomplete Injury) | 4
    ASIA D (Motor Incomplete Injury) | 0

OUTCOME MEASURES:

1. Primary Outcome: BMD of Total Hip by DXA
Description: The mean percent change in bone mineral density (BMD) of the hip after 12 months of treatment. BMD was evaluated by dual-energy X-ray absorptiometry (DXA). DXA scans measure bone density in different areas of the body using low-dose X-ray beams.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Percent change | 1.32 [-1.1 to 3.75]

2. Secondary Outcome: C-terminal Telopeptide (CTX)
Description: The mean percent change in C-terminal telopeptide (CTX) from baseline after 12 months of treatment. CTX is a bone marker found in blood serum and measures the rate of bone breakdown.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Percent change | -61.8 [-99.8 to -23.7]

3. Secondary Outcome: BMD by DXA at the Lumbar Spine
Description: The mean percent change in bone mineral density (BMD) in the lumbar spine after 12 months of treatment. BMD was evaluated by dual-energy X-ray absorptiometry (DXA). DXA scans measure bone density in different areas of the body using low-dose X-ray beams.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Percent change | 2.54 [0.17 to 4.90]

4. Secondary Outcome: Amino-terminal Propeptide of Type 1 Collagen (P1NP)
Description: The mean percent change in amino-terminal of type 1 collagen (P1NP) from baseline after 12 months of treatment. P1NP is a bone marker found in blood serum and provides information about how fast the body is making new bone.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Percent change | -51.5 [-93.8 to -9.27]

5. Secondary Outcome: Bone-specific Alkaline Phosphatase (BSAP)
Description: The mean percent change in bone-specific alkaline phosphatase (BSAP) after 12 months of treatment. BSAP is a bone marker found in blood serum and measures the rate of bone breakdown.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alendronate, Calcium, Vitamin D
Number analyzed (Participants) | 17
Percent change | -15.5 [-50.6 to 19.5]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Alendronate, Calcium, Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate, Calcium, Vitamin D (N=17)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
Sepsis (Renal and urinary disorders) | 1 (2) — Secondary to Urinary Tract Infection
Inferior Vena Cava (IVC) filter shifted (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord cysts (Nervous system disorders) | 1 (1)
Pressure sore (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate, Calcium, Vitamin D (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abscess (perineal) (Skin and subcutaneous tissue disorders) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Blood clot (Blood and lymphatic system disorders) | 1 (1)
Cold (Infections and infestations) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Cyst (Skin and subcutaneous tissue disorders) | 2 (2)
Decrease sensation (Nervous system disorders) | 1 (1) — Loss of sensation in left hand
Dizziness (Injury, poisoning and procedural complications) | 1 (1) — Lightheaded during blood draw
Eye stye (Eye disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (2)
Hernia (Gastrointestinal disorders) | 1 (1)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Endocrine disorders) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 1 (1)
Infection (MRSA) (Infections and infestations) | 1 (1)
Loose tooth (General disorders) | 1 (1)
Lower extremity fracture (Injury, poisoning and procedural complications) | 1 (1) — Distal femoral fracture
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pressure sore (Skin and subcutaneous tissue disorders) | 2 (2)
Ruptured stitches (Injury, poisoning and procedural complications) | 1 (1)
Soreness (Musculoskeletal and connective tissue disorders) | 2 (2)
Spasms (Nervous system disorders) | 1 (1)
Benign mass removal (Surgical and medical procedures) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 3 (4)
Worsened vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No